CLINICAL TRIAL: NCT07065292
Title: Investigation of the Relationship Between Plantar Sensation, Lower Extremity Position Sense, and Weight-Bearing Asymmetry With Posture, Balance, and Mobility in Individuals With Chronic Stroke
Brief Title: Plantar Sensation, Position Sense, and Weight-Bearing Asymmetry Related to Balance and Mobility Post-Stroke
Status: Recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yunus Emre Kundakçı, Assoc. Prof., Afyonkarahisar Health Sciences University
Other Study IDs: 2025/5-223
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Stroke; Sensory Impairments; Postural Control; Balance
Keywords: Chronic Stroke; Somatosensory Function; Plantar Sensation; Balance Assessment; Weight-Bearing Asymmetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine how sensory deficits and weight-bearing asymmetry affect posture, balance, and mobility in individuals with chronic stroke. The research focuses on evaluating the relationships between plantar foot sensation, lower extremity position sense, and asymmetrical weight distribution with functional abilities such as walking and postural control.

Participants will undergo non-invasive assessments, including sensation tests, mobility and balance evaluations, and postural measurements. A total of 24 individuals with chronic stroke who are receiving physiotherapy at a rehabilitation center in Konya, Türkiye, will be included.

The results of this observational, cross-sectional study may contribute to a better understanding of the sensory-motor interactions in stroke survivors and support the development of more targeted rehabilitation strategies.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability and functional impairment worldwide. Chronic stroke survivors often experience sensory deficits, particularly in the plantar surface of the foot and in lower limb proprioception. These impairments may contribute to asymmetrical weight-bearing, postural instability, and reduced mobility, all of which can negatively impact independence and quality of life.

This observational, cross-sectional study is designed to explore the associations between sensory functions (plantar sensation and lower extremity position sense), weight-bearing asymmetry, and functional outcomes including posture, balance, and walking ability. The study will be conducted on 24 individuals diagnosed with chronic stroke who are currently receiving physiotherapy as part of a personalized rehabilitation program.

All participants will be evaluated using standardized clinical assessment tools commonly employed in neurorehabilitation. These include the Semmes-Weinstein Monofilament Test for plantar sensation, a clinical position sense test for proprioception, dual-scale measurements for weight-bearing asymmetry, and functional tests such as the Postural Assessment Scale for Stroke Patients (PASS-T), Timed Up and Go Test (TUG), STREAM mobility subtests, Berg Balance Scale, Tinetti Performance-Oriented Mobility Assessment, and the Activity-Specific Balance Confidence Scale.

By identifying the relationships among sensory deficits, postural control, and functional mobility, the findings of this study may provide valuable insights for physiotherapists and rehabilitation teams in designing more effective, individualized treatment plans for chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke confirmed by a physician (via official report)
* Minimum of 6 months since stroke onset
* Aged 18 years or older
* Mini-Mental State Examination score ≥ 20
* Brunnstrom lower extremity stage ≥ 3
* Ability to complete assessments with or without walking aids
* Voluntary participation

Exclusion Criteria:

* Additional neurological, metabolic, or orthopedic conditions
* Severe vision or hearing impairments
* Modified Ashworth Score of 4 in any lower limb muscle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult individuals diagnosed with chronic stroke who are currently receiving rehabilitation services. These individuals are being treated by a licensed physiotherapist and are enrolled in individualized rehabilitation programs.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Plantar Sensation Loss (%) | Baseline
  Plantar sensation will be assessed using the Semmes Weinstein Monofilament Test. Sensory loss will be calculated as a percentage difference compared to the unaffected (healthy) side.
Lower Extremity Joint Position Sense | Baseline
  Position sense will be evaluated with the Lower Extremity Position Test. Evaluates proprioception by measuring the accuracy of toe placement on predefined distances with visual input blocked.
Weight-Bearing Asymmetry (%) | Baseline
  Weight distribution on affected and unaffected limbs will be measured using two calibrated scales. Postural symmetry index and asymmetry percentages will be calculated.

SECONDARY OUTCOMES:
Postural Assessment | Baseline
  Postural control and balance will be assessed using the Postural Assessment Scale for Stroke Patients of Turkish Version (PASS-T)
Functional Mobility | Baseline
  Timed Up and Go Test (TUG) will be used to measure the time taken to stand up, walk 3 meters, turn, return, and sit down.
Berg Balance Scale | Baseline
  It evaluates both static and dynamic balance, with total scores ranging from 0 to 56, where higher scores reflect superior balance performance.
Tinetti Balance and Gait Test | Baseline
  Tinetti Balance and Gait Test consists of two sections evaluating activities related to balance and gait. The first section includes 9 items assessing balance, while the second section comprises 7 items assessing gait. Each activity is scored based on specific observational criteria. The maximum total score is 28, with higher scores indicating better balance and gait performance. Lower scores reflect impaired balance and a higher risk of falling. Specifically, scores below 19 indicate a high risk of falls, scores between 19 and 23 indicate a moderate risk, and scores of 24 or above indicate a low risk of falling.
The Activities-specific Balance Confidence Scale | Baseline
  The Activities-specific Balance Confidence Scale is a self-reported questionnaire used to assess balance confidence in individuals with stroke. It evaluates the patient's perceived sense of safety while performing various daily activities. Each item is rated individually based on the patient's response, indicating how confident they feel about not losing their balance or falling during the activity. Scores range from 0% (no confidence at all) to 100% (complete confidence), with higher scores reflecting greater balance confidence and a lower perceived risk of falling.
Mobility & Motor Recovery | Baseline
  The Stroke Rehabilitation Assessment of Movement (STREAM) evaluates lower extremity movements and basic mobility using the final three sections of the scale. It is scored out of 35 points, with higher scores indicating better motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Kundakcı Assoc. Prof., Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Turkuaz Academy Private Education Center, Afyonkarahisar, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No